CLINICAL TRIAL: NCT03609528
Title: CamPROBE: Developing a Safer and Simple Device for Local Anaesthetic Transperineal Prostate Biopsies
Acronym: CamPROBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Vincent Gnanapragasam, Mr, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CamPROBE
Record Dates: First submitted 2018-06-06; First posted 2018-08-01 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CamPROBE biopsy method (Experimental): To be completed
  Interventions: Device: CamPROBE

INTERVENTIONS:
Device: CamPROBE — To be completed

SUMMARY:
The CamPROBE study investigates the rate of infective complications using the Cambridge Prostate Biopsy Device method of local anaesthetic transperineal prostate biopsies.

DETAILED DESCRIPTION:
The current method for diagnosing prostate cancer requires a biopsy needle to pass through the bowel wall to reach the prostate. Bacteria in the bowel inevitably enter the urinary system and blood stream. A significant number of men develop infections despite preventative antibiotics (1 in 10 develop fevers/shivers and 1-2 in 100 get a life-threatening infection). It is crucial we find a safer biopsy method for suspected prostate cancer as over 1 million rectal biopsies occur each year.

A safer alternative device was developed, performed under local anaesthetic using the transperineal route: CamPROBE (Cambridge Prostate Biopsy Device). CamPROBE biopsies are taken through the perineum (the area under the testicles), so there is no infection risk, and it's just as good at diagnosing prostate cancer. This investigation progresses from a prototype to a disposable, single use device that any UK hospital can use. The study will assess CamPROBE's ability to reduce infections from prostate biopsies and its usability as an alternative to the current standard biopsies.

Men recommended to undergo a prostate biopsy will be eligible for this multi-centre study. For each patient, the study will take approximately 30 days, consisting of: recruitment, 1 day for the procedure (replaces the standard biopsy pathway) and questionnaires on day 1, 7 and 30. This timeframe will not introduce delays in the patients' normal standard care pathway. Patients will have a transperineal biopsy with CamPROBE instead of the current transrectal method. Biopsy samples will be treated the same as standard procedure. Patients' acceptability of the procedure and complications will be measured using patient self-reported questionnaires.

ELIGIBILITY:
Inclusion Criteria:

To be included in the clinical investigation the participant must:

* Have given written informed consent to participate
* Be aged 18 years and over
* Be suitable for a prostate biopsy and clinically due to have a biopsy for diagnostic or surveillance purposes
* Be willing and able to comply with scheduled visits and completion of study questionnaires

Exclusion Criteria:

The presence of any of the following will preclude participant inclusion:

* Contraindication to a prostate biopsy
* Previous perineal or anal surgery
* Unable to lie down with legs in a stirrup for at least 45 minutes, as assessed by a clinician

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Infection | 30 days post biopsy
  Changes in incidence of infection as measured using patient self-reported Follow-Up Questionnaires and telephone assessments.

SECONDARY OUTCOMES:
Patient reported pain score | 30 days post biopsy
  Patient reported pain scores as measured using patient self-reported questionnaires.
Biological functions post biopsy | 30 days post biopsy
  Patient biological functions as measured using patient self-reported questionnaires
Patient willingness to have a repeat biopsy | 30 days post biopsy
  Patients' willingness to have a repeat biopsy as measured using patient self-reported questionnaires

OTHER OUTCOMES:
Clinician Perception | 1 day
  Clinician perception of the device and the performance of the CamPROBE assessed using Clinical Performance Assessment questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust - Addenbrooke's Hospital, Cambridge, United Kingdom